CLINICAL TRIAL: NCT02169739
Title: Pilot, Randomized, Controlled, Staggered Start, Feasibility Trial of Ischemic Preconditioning, a Promising Novel Treatment for Stroke Prevention
Brief Title: Remote Preconditioning Over Time To Empower Cerebral Tissue
Acronym: REM-PROTECT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID 19 restrictions
Sponsor: University of California, Los Angeles (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Principal Investigator, Latisha Sharma, MD, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AHA-000-376
Record Dates: First submitted 2014-06-17; First posted 2014-06-23 (Estimated); Results first posted 2021-03-10 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Ischemic Stroke; Cerebral Small Vessel Disease; Cognitive Decline
Keywords: ischemic preconditioning; remote ischemic preconditioning; ischemic stroke; white matter disease; cerebral small vessel disease; cognitive decline; leukoaraiosis; diffusion tensor imaging; white matter hyper intensity score; European scale of age-related white matter change
MeSH Terms: conditions — Ischemic Stroke; Cerebral Small Vessel Diseases; Cognitive Dysfunction; Leukoencephalopathies; Leukoaraiosis | interventions — Ischemic Preconditioning

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Medical therapy only (No Intervention): Intensive standard medical secondary prevention stroke treatment as per the recommendations of the American Heart Association/American Stroke Association national guidelines.
- Ischemic Preconditioning + Medical (Active Comparator): Patients will receive treatment with Cell Aegis remote ischemic preconditioning device once or twice daily for one year. The procedure will consist of up to four 5-minute cycles of bilateral upper extremity ischemia separated by five minutes of reperfusion. Patients will also receive intensive standard medical secondary prevention stroke treatment as per the American Heart Association/American Stroke Association national guidelines.
  Interventions: Device: Ischemic Preconditioning

INTERVENTIONS:
Device: Ischemic Preconditioning — Patients will undergo ischemic preconditioning once or twice daily for up to four 5-minutes cycles of bilateral upper extremity ischemia separated by 5-minute periods of reperfusion.
  Arms: Ischemic Preconditioning + Medical

SUMMARY:
Previous studies in animals and humans has shown that brief periods of reduced blood flow to one organ or tissue in the body can help protect other tissues from subsequent injury caused by reduced blood flow such as a stroke. This phenomenon is known as remote ischemic preconditioning and may help protect brain cells after a stroke. The investigators are studying a specific stroke type called subcortical stroke that is very common and has a high rate of recurrent stroke and cognition problems despite intensive prevention measures.

DETAILED DESCRIPTION:
In this study, the investigators will enroll 60 patients. All patients will receive best standard medical therapy for 2 years. In addition, the investigators will randomly assign 40 patients to undergo daily active remote ischemic preconditioning for 1 year, and 20 patients to 1 year of standard medical therapy followed by 1 year of daily active remote ischemic preconditioning. Patient structured interviews will be performed to assess if the treatment is well tolerated and easy for stroke patients to use. Magnetic resonance (MR) pictures of the brain will be used to determine if the active treatment stops the progression of brain injury. Cognitive tests and wireless sensor technology measures will used to learn what happens to the patient's brain and body during the active treatment.

After a subject consents to participate in the study, he/she will first participate in a study screening phase to ensure a basic level of tolerability of Remote Ischemic Conditioning (autoRIC™) device. The subject will undergo one full cycle of treatment under observation of the study team, including 4 cycles of alternating 5 minute inflation and 5 minute off periods

If the subject indicates willingness to continue receiving such treatment (screening success), she/she will enter the randomized trial phase, and be randomly allocated to the treatment or control group.

If subject indicates unwillingness to continue receiving such treatment (screening failure), he/she will not advance to the randomized phase of the trial. Screen failure subjects will be followed up with a 3-day post-device screening phone call to ensure safety and obtain information regarding any adverse events.

ELIGIBILITY:
Inclusion Criteria:

I. Clinical

1. Clinical lacunar stroke syndrome within the past 6 months
2. Absence of signs or symptoms of cortical dysfunction
3. No proximal large vessel atherosclerosis, intracranial atherosclerosis or cerebellar stroke.
4. No major cardioembolic source requiring anticoagulation or other specific therapy

II. Imaging

1. Magnetic Resonance Imaging (MRI) presence of a small subcortical ischemic, any 1 or more of:

   1. Diffusion-weighted imaging (DWI) lesion < 2.0cm in size at largest dimension and corresponding to the clinical syndrome.
   2. Well delineated focal hyperintensity <2.0 cm in size at largest dimension (including rostro-caudal extent) on FLAIR or T2 and clearly corresponding to the clinical syndrome. If other focal hyperintensities are present, the case will be discussed with the principal investigator prior to randomization
   3. Multiple (at least 2) hypointense lesions of size 0.3-1.5 cm at largest dimension (including rostro-caudal extent) only in the cerebral hemispheres on FLAIR or T1 in patients whose qualifying event is clinically hemispheric
   4. Well delinated hypointense lesion <1.5 cm in size at the largest dimension (including rostro-caudal extent) on FLAIR or T1 corresponding to the clinical syndrome. MRI must be done at least 1 months after the qualifying stroke
2. Absence of cortical stroke and large (> 1.5cm) subcortical stroke, recent or remote
3. White matter hyperintensity score of 2 (moderate) or 3 (severe) on the European Scale of Age-Related White Matter Change
4. Absence of cerebral amyloid antipathy (CAA) as per Boston Criteria.

Exclusion Criteria:

1. Disabling stroke (Rankin Scale ≥4)
2. Previous intracranial hemorrhage (excluding traumatic) or hemorrhagic stroke
3. Age under 40 years
4. High risk of bleeding (e.g. recurrent GI or GU bleeding, active peptic ulcer disease, etc.)
5. Anticipated requirement for long term use of anticoagulants (e.g. recurrent deep venous thrombosis (DVT)
6. Prior cortical or retinal stroke (diagnosed either clinically or by neuroimaging), or other prior cortical or retinal transient ischemic attack (TIA)
7. Prior ipsilateral carotid endarterectomy
8. Impaired renal function: estimated GFR <40
9. Intolerance or contraindications to aspirin or clopidogrel (including thrombocytopenia, prolonged INR)
10. Mini Mental Status Exam score < 24 (adjusted for age and education)
11. Medical contraindication to MRI
12. Pregnancy or women of child-bearing age who are not following an effective method of contraception
13. Pre-existing neurologic, psychiatric, or advanced systemic disease that would confound the neurological or functional outcome evaluations
14. SBP <90 or > 200
15. Known history of limb vascular disease, limb vascular bypass surgery, or limb deep venous thrombosis
16. Prisoners
17. Homeless individuals
18. Patient unable to give informed consent and no available legally authorized representative to provide informed consent
19. Patient unlikely to be compliant with therapy/ unwilling to return for follow up visits
20. Concurrent participation in another study with investigational drug or device treatment
21. Other likely specific cause of stroke (e.g. dissection, vasculitis, prothrombotic diathesis, drug abuse)

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2020-03 (Actual); Study Completion 2020-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Latisha K Sharma, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California Los Angeles UCLA, Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Ischemic Preconditioning + Medical: Treatment with Cell Aegis remote ischemic preconditioning device once or twice daily for one year, consisting of up to four 5-minute cycles of bilateral upper extremity ischemia separated by five minutes of reperfusion. Patients received intensive standard medical secondary prevention stroke treatment as per the American Heart Association/American Stroke Association national guidelines.
Period: Overall Study
Arm/Group | Medical Therapy Only | Ischemic Preconditioning + Medical
Started | 2 | 4
Completed | 2 | 0
Not Completed | 0 | 4
Not completed — Lost to Follow-up | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Medical Therapy Only | Ischemic Preconditioning + Medical | Total
Number analyzed (Participants) | 2 | 4 | 6
Age, Continuous [Mean (Full Range); unit: years] | 74 [73 to 75] | 63.7 [52 to 71] | 67.1 [52 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 1 | 4 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 4 | 6
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 1 | 1 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Duration of Adherence to Ischemic Preconditioning Procedure
Time Frame: 12 months
Population: The medical intervention arm did not undergo ischemic preconditioning
Measure: Median (Full Range); unit: Months
Arm/Group | Ischemic Preconditioning + Medical
Number analyzed (Participants) | 4
Months | 3 [1 to 3]

2. Secondary Outcome: Limb Ischemia as Assessed by the Preconditioning Device
Time Frame: 12 months
Population: Data were not collected since no participants reached the 12-month follow-up
Arm/Group | Medical Therapy Only | Ischemic Preconditioning + Medical
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Patient Self-reported Comfort-discomfort on a Scale of 1-5, With Lowest Score = "Very Comfortable" and 5 = "Very Uncomfortable"
Time Frame: 12 months
Population: Data were not collected since no participants reached the 12-month follow-up
Arm/Group | Medical Therapy Only | Ischemic Preconditioning + Medical
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Medical Therapy Only | Ischemic Preconditioning + Medical
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/4
Other Adverse Events (participants affected / at risk) | 0/2 | 0/4

LIMITATIONS AND CAVEATS:
We faced recruitment challenges over the course of the study. Many patients declined enrollment due to the 12-month time commitment of the study. We faced tolerability and compliance concerns with the few patients enrolled in the study. Despite our efforts, early termination of the trial led to small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-08): https://cdn.clinicaltrials.gov/large-docs/39/NCT02169739/Prot_SAP_000.pdf